CLINICAL TRIAL: NCT04171167
Title: The Causal Relation of Nasal Nitric Oxide Levels to the Severity of Chronic Rhinosinusitis and Its Inflammatory Phenotype
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R17011
Record Dates: First submitted 2018-10-23; First posted 2019-11-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Nasal nitric oxide; Nitric oxide metabolites
MeSH Terms: conditions — Disease | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Frequently treated acute rhino sinusitis (Active Comparator): Does not meet the European position paper criteria of CRS: asymptomatic periods in between and no objective findings when entering the study.
  Interventions: Drug: Fluticasone Propionate
- CRSsNP (Active Comparator): Meets the European position paper criteria of CRS. Zinreich modification of Lund-Mackey scoringing: Opacification score < 21 and obstruction score 0-8. No visible nasal polyps in endoscopy
  Interventions: Drug: Fluticasone Propionate
- Severe CRSsNP and CRSwNP (Active Comparator): Meets the European position paper criteria of CRS and not included in the first two groups.
  Interventions: Drug: Fluticasone Propionate
- Healthy volunteers (No Intervention): No nasal symptoms or complaints. No interventions done.

INTERVENTIONS:
Drug: Fluticasone Propionate — three visits: 0, after washout, after FP usage
  Arms: CRSsNP; Frequently treated acute rhino sinusitis; Severe CRSsNP and CRSwNP

SUMMARY:
Nitric oxide (NO) reflects changes in inflammatory state of the airways. In pulmonology fractional exhaled nitric oxide concentration (FeNO) has been linked to eosinophilic asthma and is used to guide overall disease control. The measurement of nasal nitric oxide (nNO) may reflect the disease burden and inflammatory phenotype of the paranasal sinuses.

The aim of our study is to evaluate the relation of chronic rhino sinusitis (CRS) severity and inflammatory status to nNO, maxillary sinus NO, nitrite, nitrate and cone beam computed tomography (CBCT).

Three groups (22 patients in each) of referred patients and and 22 healthy volunteers are recruited. Patients are grouped according to the CBCT score and viewed three times in 4-6 weeks intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate in the study
* Patients who are referred to ENT clinic due to chronic rhinosinusitis (EPOS criteria) or repeatedly diagnosed and treated acute rhinosinusitis

Exclusion Criteria:

* Endoscopic sinus surgery operation previously
* Septal deviation that would need an operation to correct the air flow
* Other severe disease that could pose a risk for the patient during the measurements based on the judgement of the treating physician
* Pregnancy or breastfeeding
* Allergy to used medications
* Inability to co-operate or to tolerate manipulation of the nose

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Nasal nitric oxide levels | Change between visit: 0, +5 weeks, +10weeks
  Gaseous nitric oxide is measured nasal cavity and maxillary sinuses using EcoMedics CLD 88p analyser (ppb). Procedure according to ERS protocol.
Nitric oxide metabolite (nitrate, nitrite) levels | Change between visit: 0, +5 weeks, +10weeks
  NO production is determined from saline lavage of nasal cavity and maxillary sinus by measuring the accumulation of nitrite, a stable metabolite of NO in aqueous milieu, by the Griess reaction

SECONDARY OUTCOMES:
CBCT (Zinreich modified Lund-Mackay) scoring | Change between visit: 0, +5 weeks, +10weeks
  A routine high resolution cone beam computed tomography (CBCT) is done to evaluate the initial status of the patients nose and repeated (with ultra-low-dose protocol) at every visit to demonstrate the the current state.
  Opasification score scale 0-5, max. 50 and obstruction score 0-1 (0,5 steps), max. 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided